CLINICAL TRIAL: NCT06016387
Title: Tucatinib, Trastuzumab and Capecitabine With Brain and/or Spinal Radiotherapy (XRT) in Patients With HER2+ Metastatic Breast Cancer and Leptomeningeal Disease: A Multi-centre Phase II, Single Arm Feasibility Study
Brief Title: Tucatinib With Brain and/or Spinal XRT in Patients With HER2+ Metastatic Breast Cancer and LMD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Biocon Biologics (Unknown); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLIMB-LMD
Record Dates: First submitted 2023-08-18; First posted 2023-08-29 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-01

CONDITIONS: HER2-positive Breast Cancer; LMD
Keywords: HER2+; Breast Cancer; Leptomeningeal disease; Tucanitib; CLIMB-LMD; HER2 CLIMB LMD; CLIMB LMD HER2+
MeSH Terms: conditions — Breast Neoplasms; Meningeal Neoplasms | interventions — tucatinib; Trastuzumab; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tucatinib, Transtuzumab, Capecitabine (Experimental): Tucatinib, Trastuzumab and Capecitabine With Brain and/or Spinal Radiotherapy (XRT) in Patients With HER2+ Metastatic Breast Cancer and Leptomeningeal Disease.
  Interventions: Drug: Tucatinib 150 MG; Drug: Trastuzumab; Drug: Capecitabine; Radiation: Brain & Spinal Radiation

INTERVENTIONS:
Drug: Tucatinib 150 MG — Tucatinib is a potent, selective, adenosine triphosphate-competitive small-molecule inhibitor of the receptor tyrosine kinase HER2. The molecular formula for tubatinib is C26H24N8O2 and it has a molecular weight of 480.52 g/mol.
  Other Names: Tukysa
Drug: Trastuzumab — MYL-1401O contains the active substance trastuzumab, which is an IgG1 monoclonal antibody. The molecular size of the intact molecule is around 148 kDa.
  Each vial of MYL-1401O contains 150 mg of lyophilized proposed active biosimilar substance trastuzumab as well as 3.36 mg L-Histidine Hydrochloride, 2.16 mg L-Histidine, 115.2 mg sorbitol and 33.6 mg PEG-3350 (Macrogol 3350). Sorbitol and PEG-3350 substitute the α- trehalose dehydrate and polysorbate-20, which are used as excipients in the EU-approved and US-licensed Herceptin formulations.
Drug: Capecitabine — Capecitabine is a tumour-activated antineoplastic agent (antimetabolite). The molecular formula for capecitabine is C15H22FN3O6 and has a molecular weight of 359.35 g/mol.
Radiation: Brain & Spinal Radiation — Brain & Spinal XRT is a treatment for patients with HER2+ metastatic breast cancer and leptomeningeal disease,
  Other Names: Brain & Spinal XRT

SUMMARY:
The proposed study will evaluate the safety and efficacy of XRT followed by systemic therapy among patients with HER2+ metastatic breast cancer and LMD

DETAILED DESCRIPTION:
Breast cancer is the most common cancer among women worldwide, and the second leading cause of brain metastases (BrM). Despite recent treatment advances, the prognosis of patients with breast cancer BrM remains poor, and the prognosis among those with leptomeningeal disease (LMD) is particularly dire with a median survival of only 2-4 months.

Patients with HER2+ metastatic breast cancer have a high life-time risk of central nervous system (CNS) metastases, with an approximately 50% lifetime risk. Although the cause of death among patients with breast cancer BrM is challenging to ascertain, approximately 50% of patients with HER2+ BrM are thought to die from central nervous system (CNS) disease involvement. Among patients with LMD specifically, the cause of death is most commonly related to CNS disease.

In an analysis of 430 patients (96 of whom had breast cancer) treated for LMD in the National Cancer Database between 2005 and 2014, those patients treated with chemotherapy plus radiotherapy had a longer median overall survival of 5 months (3.5 - 6.5 months) compared to patients treated with XRT or chemotherapy alone. In addition, a majority (n=18/26, 69%) of observational studies irrespective of primary tumor site have shown an "improvement or likely improvement" in survival with the use of XRT for LMD, either alone or in combination with systemic therapy. Hence, this proposed study will evaluate the safety and efficacy of XRT followed by systemic therapy (which is considered standard of care) among patients with HER2+ metastatic breast cancer and LMD.

ELIGIBILITY:
Inclusion Criteria: Phase 1

1. Men or women with HER2+* metastatic breast cancer. *HER2+ status will be defined in accordance with ASCO-CAP 2018 guidelines, and can be diagnosed at any time prior to enrolment;
2. Evidence of LMD* in the brain and/or spine (either positive cerebral spinal fluid cytology and/or magnetic resonance imaging evidence of LMD). Measurable disease in the central nervous system is not required. * The diagnosis of LMD can occur at any time prior to enrolment;
3. Age 18+ at time of consent;
4. ECOG ≤ 2;
5. More than 14 days or 5 half-lives from the last dose of any experimental agent is required, whichever is greater;
6. All toxicity related to prior cancer therapies must have resolved to ≤ Grade 1 prior to enrollment, except for alopecia; neuropathy, must have resolved to ≤ Grade 2.

Phase 2: Inclusion Criteria

1. Left ventricular ejection fraction (LVEF) must be within institutional limits of normal as assessed by ECHO or MUGA documented within 2 weeks prior to starting systemic therapy on the study;
2. Adequate hematologic, liver, and renal function within 2 weeks prior to phase 2 enrollment, as follows:

   1. Hemoglobin ≥ 9 g/dL
   2. ANC ≥ 1 x109/L
   3. Platelets ≥ 100 x109/L
   4. Total bilirubin ≤ 1.5 X upper limit of normal (ULN)
   5. AST and ALT ≤ 2.5X ULN
   6. International normalized ratio (INR) and activated partial thromboplastin time (aPTT) ≤ 1.5 X ULN
   7. Creatinine clearance (CrCL) ≥ 50 mL/min
3. The last dose of prior therapy must have been completed 14 days prior to study enrollment. Prior chemotherapy, immunotherapy, endocrine therapy, targeted therapy and experimental agents are allowed (including prior use of trastuzumab or other antibody-based therapy). Prior use of capecitabine either alone or in combination with other HER2-targeted therapies (including other tyrosine kinase inhibitors) is permitted;

Exclusion Criteria: Phase 1

1. Prior WBRT for brain metastases (prior stereotactic radiosurgery for parenchymal CNS metastases received <7 days prior to consent );
2. Prior therapy specifically directed at LMD, including prior radiotherapy or systemic therapy;
3. Inability to comply with MRI-based surveillance of CNS disease;
4. Inability to swallow pills or any significant gastrointestinal diseases such as inflammatory bowel disease who suffer from uncontrolled diarrhea (based on the investigator's assessment),, which would preclude adequate absorption of oral medications;
5. Diagnosed with Hereditary fructose intolerance;
6. Diagnosed with Gilbert's disease;
7. Prior history of other cancer (except non melanoma skin, cervical intraepithelial neoplasia) with evidence of disease within the last 5 years;
8. Prior use of tucatinib at any time prior to enrollment.
9. Hypersensitivity to any of the active substances in tucatinib, trastuzumab, or capecitabine.

Phase 2:

1. Currently pregnant or breastfeeding;
2. Use of a strong cytochrome P450 (CYP)2C8 inhibitor within 5 half-lives of the inhibitor or use of a strong CYP3A4 or CYP2C8 inducer within 5 days prior to the first dose of systemic therapy (see Appendix C and D);
3. Myocardial infarction or unstable angina within 6 months prior to the first dose of systemic therapy.
4. Blood product transfusions in order to meet eligibility criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-11-25 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-10-05 (Estimated)

PRIMARY OUTCOMES:
Survival status from the start of XRT • Survival status from the start of XRT | From date of baseline until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  To assess overall survival (OS) from the start of XRT.

SECONDARY OUTCOMES:
Time to CNS progression from the start of XRT | From date of baseline until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  To determine the time for CNS symptoms progresses from start of XRT in the proposed patient population after completion of brain and/or spinal XRT.
  To determine the efficacy of tucatinib plus trastuzumab and capecitabine for the treatment of patients with HER2+ breast cancer and leptomeningeal metastases (LMD).
Safety and tolerability (CTCAE v.5.0) | From date of baseline until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  To determine the safety & tolerability of systemic therapy (tucatinib, trastuzumab and capecitabine) in the proposed patient population after completion of brain and/or spinal XRT.
  To determine the efficacy of tucatinib plus trastuzumab and capecitabine for the treatment of patients with HER2+ breast cancer and leptomeningeal metastases (LMD).
Progression free survival from the start of XRT | From date of baseline until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  To determine progression from the start of XRT in the proposed patient population after completion of brain and/or spinal XRT.
  To determine the efficacy of tucatinib plus trastuzumab and capecitabine for the treatment of patients with HER2+ breast cancer and leptomeningeal metastases (LMD).
CNS specific objective response (RANO-BM) | Every 6 weeks through study completion, an average of 5 years
  To determine the CNS objective response in the proposed patient population after completion of brain and/or spinal XRT.
  To determine the efficacy of tucatinib plus trastuzumab and capecitabine for the treatment of patients with HER2+ breast cancer and leptomeningeal metastases (LMD).
Extracranial objective response (RECIST v1.1) | Every 6 weeks through study completion, an average of 5 years
  To determine the extracranial objective response in the proposed patient population after completion of brain and/or spinal XRT.
  To determine the efficacy of tucatinib plus trastuzumab and capecitabine for the treatment of patients with HER2+ breast cancer and leptomeningeal metastases (LMD).
Neurologic-specific QoL (FACT-BR version 4) | Pre-treatment, at the start of Cycle 3 (Cycle 3 Day 1, +/- 7 days) and at the Safety Visit
  To determine the neurologic-specific QoL's in the proposed patient population after completion of brain and/or spinal XRT.
  To determine the efficacy of tucatinib plus trastuzumab and capecitabine for the treatment of patients with HER2+ breast cancer and leptomeningeal metastases (LMD).
Overall QoL (EORTC QLQ-C30 version 3) | Pre-treatment, at the start of Cycle 3 (Cycle 3 Day 1, +/- 7 days) and at the Safety Visit
  To determine the Overall QoL in the proposed patient population after completion of brain and/or spinal XRT.
  To determine the efficacy of tucatinib plus trastuzumab and capecitabine for the treatment of patients with HER2+ breast cancer and leptomeningeal metastases (LMD).

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - The Ottawa Hospital, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No
The Aggregate data will be presented and/or published. The IPD will not be available keeping patients privacy in mind.